CLINICAL TRIAL: NCT04231032
Title: Paced Dyssynchrony and Myocardial Perfusion IN apiCal Hcm
Acronym: PINCHcm
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit to target
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: V1.2_25 08 21
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Apical hypertrophic cardiomyopathy; Pacemaker; Perfusion
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Apical Hypertrophic Cardiomyopathy

STUDY DESIGN:
Intervention Model Description: Double-blind, randomised, cross-over design
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active ventricular pacing (Active Comparator): Asynchronous dual chamber pacing (DOO mode) at a heart rate just higher than that expected to be achieved with adenosine infusion (same rate in each arm)
  Interventions: Other: Asynchronous dual chamber pacing (DOO) with paced ventricular activation
- Back-up ventricular pacing (Placebo Comparator): Asynchronous atrial pacing with intrinsic ventricular activation (AOO mode) at a heart rate just higher than that expected to be achieved with adenosine infusion (same rate in each arm)
  Interventions: Other: Asynchronous atrial pacing (AOO) with intrinsic ventricular activation

INTERVENTIONS:
Other: Asynchronous dual chamber pacing (DOO) with paced ventricular activation — Alteration of the participant's existing pacemaker mode to either paced or intrinsic ventricular activation (in an order based upon randomisation).
  Arms: Active ventricular pacing
Other: Asynchronous atrial pacing (AOO) with intrinsic ventricular activation — Alteration of the participant's existing pacemaker mode to either paced or intrinsic ventricular activation (in an order based upon randomisation).
  Arms: Back-up ventricular pacing

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is the most common inherited heart disease. A relatively common subgroup of HCM patients have apical HCM - a type of heart muscle disease that causes abnormal muscle thickening towards the tip (apex) of the heart. This can impair the heart's own blood flow through the thickened heart muscle. We think this is one of the causes for symptoms such as shortness of breath and chest pain. If medications are ineffective at treating symptoms, there are few further options available, limited to invasive heart surgery.

This study aims to determine if it is possible to improve the blood flow within by altering the settings of patients' permanent pacemakers, dynamic microvascular obstruction is an important cause of perfusion abnormalities in HCM and whether introducing localized dyssynchrony with ventricular pacing improves this. This phased study will include patients with apical HCM that already have implanted pacemaker devices to remove risks associated with device implantation.

The study may provide insights into novel mechanisms for symptoms in HCM and provide new methods for treating a patient group in whom therapeutic options can be extremely limited.

DETAILED DESCRIPTION:
The treatments for people with apical HCM and symptoms are limited but include medicines. The use of a pacemaker in this situation is an experimental treatment which has not yet been fully explored. We believe symptoms are linked with abnormalities in blood flow through the heart muscle at the tip / apex of the heart and wish to see if using a pacemaker can improve such abnormalities. We want to test if this treatment works using a clinical trial to help us decide whether this is a viable treatment option that may be offered to other patients with the condition. The null hypothesis states that there will be no difference in blood flow through the heart muscle with pacing. The alternative hypothesis states that there will be a significant difference in blood flow through the heart muscle with pacing. This was chosen based upon our current knowledge that abnormal blood flow in the heart muscle in apical HCM is linked with abnormal squeeze at the apex / tip and symptoms. Echocardiography pilot data has demonstrated a reduction in squeeze at the apex of the heart when using the pacemaker to cause the heart muscle to contract in a different way.

Our alternative hypothesis therefore is that we can use the pacemaker to reduce squeeze at the apex and improve blood flow through the heart muscle. This is a single centre, prospective pilot study. Because data on acute changes in perfusion with pacing in apical HCM are extremely limited, the most ethical methodology is to perform a two-phase study. Phase A of the study assesses acute changes in blood flow through the heart muscle during different pacemaker settings (active and back-up), looking for potential efficacy of the intervention. Secondary outcomes of Phase A include recruitment rate and proportion of patients willing to proceed to Phase B. Phase B of the study consists of entering those same patients into a randomised double-blind cross-over 6-month follow-up pilot to collect baseline statistical data and assess acceptability of study protocol to design a future study. Here, assessment of further secondary outcomes will allow establishment of baseline statistical data for the design of an outcomes-based clinical trial. Patients will only be entered into phase B of the study if an improvement is seen in myocardial perfusion with pacing during phase A.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, >18 years.
2. HCM patients with apical HCM defined as apical hypertrophy with apical LV systolic obliteration and the presence of characteristic ECG changes. Participants with a mixed cardiac phenotype will be considered if they also meet these criteria and do not have resting outflow tract obstruction.
3. A programmable intracardiac pacing device with a right atrial lead and an apically / low septal located right ventricular lead.
4. Willing and able to provide informed consent.

Exclusion Criteria:

1. Outflow tract obstruction >50 mmHg at rest due to systolic anterior mitral movement.
2. Evidence of high-grade heart block.
3. Moderate or severe primary valvular disease.
4. Unrevascularised, known, significant coronary disease: the significance of any known coronary disease will be determined after discussion with an independent clinician.
5. Atrial fibrillation at the time of randomisation.
6. Inability to undergo CMR with adenosine stress and gadolinium contrast imaging.
7. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion mapping | Acute changes during the CMR scan on Visit 1 (day 1)
  Percentage change in regional myocardial perfusion between baseline and pacing measured using myocardial blood flow (MBF) mapping at Cardiovascular Magnetic Resonance (CMR) imaging.

SECONDARY OUTCOMES:
Proportion successfully completing the CMR scan with interpretable images. | After all visit 1 completed (within 6 months)
  Number of participants whose perfusion imaging is readable
Myocardial contractility via CMR | Acute changes during the CMR scan on Visit 1 (day 1)
  Alterations in regional and global myocardial contractility and relaxation measured by cardiac magnetic resonance imaging.
Myocardial contractility via echocardiography | Acute changes during the echocardiogram scan on Visit 1 (day 1)
  Alterations in regional and global myocardial contractility and relaxation measured by echocardiography.
Proportion unwilling to proceed to Phase B. | After all visit 1 completed (within 6 months).
  Proportion of participants who are unwilling to proceed to Phase B.
Recruitment rate. | 12 months.
  The rate at which participants are recruited into the study.
Exercise performance on Bruce protocol treadmill exercise tolerance test (ETT) | 3 and 6 months
  Time in minutes on the Bruce protocol ETT with active or back-up ventricular pacing.
Exercise performance on 6-minute walk test (6MWT). | 3 and 6 months
  Distance walked in metres during 6-minute walk test (6MWT) with active or back-up ventricular pacing.
Seattle Angina Questionnaire score | 3 and 6 months
  Seattle Angina Questionnaire score with active or back-up ventricular pacing. The SAQ is a self-administered, disease-specific measure for patients with CAD that is valid, reproducible, and sensitive to clinical change. This instrument was developed and validated by John Spertus, Director of Cardiovascular Education and Outcomes Research at the Mid America Heart Institute and Professor of Medicine at the University of Missouri - Kansas City. The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).
Short-form 36 (SF36) questionnaire score | 3 and 6 months
  SF36 Questionnaire score with active or back-up ventricular pacing. The RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Euroqol 5 domain 5 level (EQ5D-5L) questionnaire score | 3 and 6 months
  EQ5D-5L Questionnaire score with active or back-up ventricular pacing. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
New York Heart Association (NYHA) classification. | 3 and 6 months
  New York Heart Association (NYHA) classification with active or back-up ventricular pacing. The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
Proportion of accidental un-blinding. | 12 months.
  Proportion of participants who are accidentally un-blinded to their pacemaker settings during follow-up.
Proportion of patients requesting cross-over due to symptoms. | 12 months.
  Proportion of patients requesting cross-over due to symptoms during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Saidi A Mohiddin, MBChBFRCPMD, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Heart Centre, London, Thames, United Kingdom

IPD SHARING:
Plan to Share IPD: No